CLINICAL TRIAL: NCT06563375
Title: Phase 1 Dose Escalation and Dose Expansion Trial of NP-101 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novatek Pharmaceuticals, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0500; NCI-2024-06908 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental)
  Interventions: Drug: NP-101
- Dose Expansion (Experimental)
  Interventions: Drug: NP-101

INTERVENTIONS:
Drug: NP-101 — Given by mouth

SUMMARY:
To evaluate the safety and preliminary efficacy of NP-101 in patients with solid tumors.

DETAILED DESCRIPTION:
Primary Objective:

To determine the safety and tolerability of NP-101 in patients with solid tumors.

Secondary Objective:

To determine the preliminary antitumor activity of NP-101. Although the clinical benefit of NP-101 has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit and thus, the patient will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability.

Exploratory Objectives:

To evaluate immune-related markers of response and resistance to NP-101. To bank blood samples for future pharmacokinetic (PK) analyses of NP-101.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years.
2. Must be willing and able to provide informed consent.
3. Ability to comply with the study protocol, in the investigator's judgment.
4. Histologically documented advanced or metastatic solid tumor that has relapsed or progressed following local standard treatments that are known to prolong survival, or for which no standard treatment is available.
5. For dose escalation, patients can have evaluable or measurable disease. For dose expansion, patients must have measurable disease per the RECIST v1.1 (Appendix 1).
6. Eastern Cooperative Oncology Group performance status of 0 or 1 (Appendix 2).
7. Life expectancy 3 months.
8. Adequate organ and marrow function as defined below within 28 days of study treatment initiation:

   * Hemoglobin >9.0 g/dL
   * Absolute neutrophil count ≥1500/mL
   * Platelets ≥100,000/mL
   * Total bilirubin ≤1.5 institutional upper limit of normal (ULN). Documented Gilbert syndrome is allowed if total bilirubin is ≤3 × ULN.
   * Aspartate transaminase/ALT ≤3 × institutional ULN.
   * Creatinine clearance ≥60 mL/min.
   * For patients not receiving therapeutic anticoagulation: international normalized ratio or activated partial thromboplastin time ≤1.5 × ULN. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
9. Left ventricular ejection fraction ≥50%.

9. Patients must have adequate washout from prior therapy at the time of study treatment initiation: 4 weeks from major surgery; 4 weeks from antibody-based therapy; 2 weeks or 5 half-lives (whichever is shorter) from any targeted therapy or small molecule therapy; 3 weeks or 5 half-lives (whichever is shorter) from chemotherapy or 6 weeks in the case of certain therapies (e.g., extensive radiotherapy, mitomycin C, and nitrosoureas); and 4 weeks from radiation therapy. Palliative radiotherapy is permitted for a preexisting lesion, provided it does not interfere with the assessment of tumor target lesions (e.g., the lesion to be irradiated must not be a site of measurable disease).

10. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational agent are eligible for this study.

Women of childbearing potential (WOCBP) must agree to follow the contraception guidelines in Appendix 3 during the study treatment period and for at least 60 days after the last dose of study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a post-menopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Female patients who become pregnant will be taken off study.

12. Male patients of childbearing potential must agree to follow the contraception guidelines in Appendix 3 during the study treatment period and for at least 60 days after the last dose of study treatment.

13. WOCBP must have a negative serum pregnancy test result within 3 days of study treatment initiation.

14. Willing to undergo mandatory tumor biopsy and blood collections as required by the study.

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug.
2. Unresolved toxicities from prior therapy (defined as having not resolved to NCI CTCAE v.5.0 Grade ≤1 or baseline). Exceptions include endocrinopathies from prior therapy or disease and successfully treated (such as hypothyroidism, diabetes mellitus), alopecia, vitiligo, and Grade ≤2 peripheral neuropathy. Patients may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to Grade >2 for at least 3 months prior to Cycle 1, Day 1 and managed with standard of care treatment) that the investigator deems related to previous toxicities from prior immunotherapy treatment.
3. Patients who are receiving any other investigational agents.
4. Unable to swallow and retain oral medications.
5. Gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
6. Known positive status for HIV infection.
7. Known active hepatitis B virus or HCV infection.
8. Brain or leptomeningeal metastases.
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
10. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the investigator.
11. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal).
12. Active infection requiring systemic antimicrobial treatment (including antibiotics, antifungals, and antiviral agents).
13. Clinically significant cardiovascular disease within 12 months prior to enrollment, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebrovascular event, or cardiac arrhythmia associated with hemodynamic instability. NOTE: medically controlled arrhythmia would be permitted.
14. Pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT06563375/ICF_000.pdf